CLINICAL TRIAL: NCT05293002
Title: Belgian Study to Assess the Efficacy and Safety of the RESTORER Iliac Stent System for the Treatment of Aorto-iliac Lesions (TASC A, B, C and D).
Brief Title: Belgian Study to Assess the Efficacy and Safety of the RESTORER Iliac Stent for Treatment of Aorto-iliac Lesions.
Acronym: BARISTA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ID3 Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BARISTA protocol v3.0 20230405
Record Dates: First submitted 2022-01-19; First posted 2022-03-23 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: All patients will receive the Restorer stent of iVascular according to the IFU. Prospective, single-arm, multicentre, physician-initiated clinical study to assess the safety and efficacy of the study device during a two year FU period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Restorer Iliac Stent System (Experimental): RESTORER Iliac Stent system for the treatment of Aorto-iliac lesions (TASC A, B, C and D) according to IFU
  Interventions: Device: Restorer Iliac Stent System

INTERVENTIONS:
Device: Restorer Iliac Stent System — Not applicable (only one intervention)

SUMMARY:
The BARISTA study tests the safety and efficacy of the Restorer stent from the company iVascular. This stent is a medical device that is already approved for use in Europe, to treat stenotic (narrowed) iliac arteries. 200 Belgian patients from 13 different hospitals will be included in this study. Patients will be medically monitored for 2 years from the day of the study procedure. The treatment of the stenotic iliac arteries will be according to the standard of care, using the Restorer stent. This endovascular treatment consists of introducing the necessary materials in the blood vessels by a puncture in the groin under general or local anaesthesia, after which a thin plastic tube will be inserted into the femoral artery through the puncture site, until the stenotic iliac artery is reached. Medical imaging is done by angiography. The stenotic/occluded section of the artery will first be dilated by inserting and inflating a balloon. Next, the Restorer stent will be placed and, if necessary, another balloon may be inserted and inflated to allow the stent to fit nicely to the vessel wall and optimise the result. As per standard of care, follow-up will be done in the hospital after 1, 6, 12, and 24 months. During these visits, an ultrasound scan of the treated artery will be taken to evaluate the patency of the blood vessel. Also, two short questionnaires will be completed asking about the quality of life and walking difficulties. The use of medication will be recorded. If adverse events are experienced, they will be reported.

DETAILED DESCRIPTION:
Prospective, single-arm, multicentre, physician-initiated clinical study to assess the long-term (up to 24 months) safety and efficacy of the RESTORER peripheral stent system (iVascular) for the treatment of iliac lesions in 200 subjects, in a controlled clinical setting post CE-certification when used according to the IFU with focus on the treatment of complex TASC A, B, C and D Aorto-iliac lesions. The primary endpoint of the study is freedom of any TLR, major amputation or restenosis (defined as significant stenosis on duplex ultrasound (>50%, systolic velocity ratio greater than 2.4) within 12 months. Secondary endpoints are: technical success during procedure, and during the follow-up period: primary patency, stent graft occlusion rate, ABI, freedom from target lesion revascularization, clinical success (improvement of Rutherford classification), change in walking impairment questionnaire, change in quality of life questionnaire, freedom from above-the-ankle target limb amputation, and mortality. A subanalysis will be done to compare the results using the TASC classification, lesion location (AIE, AIC, bilateral, kissing configuration), gender, diabetes mellitus and Rutherford in terms of patency, frequency of TLR and clinical outcome at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria: 1. Males or non-pregnant females ≥ 18 years of age at the time of consent. Females of childbearing potentials have a negative pregnancy test <7 days before the procedure and are willing to use a reliable method of birth control for the duration of study participation. Female participants will be exempted from this requirement in case they are sterile, infertile or have been post-menopausal for at least 12 months.

2. Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study.

3. Patient presenting with a stenotic or occlusive lesion at the Aorto-iliac arteries suitable for stenting with the Restorer stent (iVascular) (on indication for primary stenting, based on the discretion of the investigator). This lesion is corresponding to the CE-mark indications/contra-indications and according to the current medical guidelines for minimally invasive peripheral interventions.

4. Estimated life expectancy ≥ 2 years. 5. Patient presenting a score from 2 to 4 following Rutherford classification. 6. Patient is willing to comply with specified follow-up evaluations at the specified times for the duration of the study.

7. The target lesion has angiographic evidence of stenosis or restenosis >50% or occlusion which can be passed with standard guidewire manipulation.

8. There is angiographic evidence of a patent Common and Deep Femoral Artery.

-

Exclusion Criteria: 1. Patients with a history of coagulation disorders, 2. Presence of an aneurysm immediately adjacent of the site of stent implantation, 3. Extension of more than 1cm in distal aorta, 4. Extension into CFA, 5. Fresh thrombus formation, 6. Acute limb ischemia, defined as symptom onset during less than 14 days prior to the index procedure, 7. Any systemic infection or immunocompromised state. Patients with an ascending infection/deep foot infection or abscess/white blood count (WBC)≥12.000/or febrile state or CRP>5mg/L, 8. Existing stent implant in the target vessel, 9. Use of alternative therapies: atherectomy, cutting/scoring balloons, laser, … 10. Known coagulopathy, hypercoagulable state, bleeding diathesis, other blood disorder, or a platelet count less than 80.000/µL or greater than 500.000/µL, 11. Any subject in which antiplatelet, anticoagulant or thrombolytic therapy is contraindicated, 12. Known hypersensitivity or contraindication to the stent material (CoCr L605), 13. Has other comorbidities that, in the opinion of the investigator, would preclude them from receiving this treatment and/or participating in study-required follow-up, 14. Known hypersensitivity or allergy to contrast agents that cannot be medically managed, 15. Inadequate inflow lesion treatment (>30% residual stenosis), 16. Subject has IFU listed contraindication(s).

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from TLR | 12 months
  Freedom from any Target Lesion Revascularization (TLR) at 12 months
Freedom from major amputation | 12 months
  Freedom from amputation above the ankle
Freedom from restenosis | 12 months
  No significant stenosis on duplex ultrasound (>50% stenosis or systolic velocity ratio greater than 2.4)

SECONDARY OUTCOMES:
Technical success | 1 month
  final residual angiographic stenosis <30%
Primary patency rate | 6, 12, and 24 months
  lack of restenosis and no need for reintervention of the target lesion
Stent graft occlusion rate | 1, 6, 12, and 24 months
  Presence or absence of occlusion
ABI | 6, 12, and 24 months
  comparison of Ankle Brachial Index at follow-up compared to baseline ABI
Freedom from Target Lesion Revascularization | 12 and 24 months
  freedom from repeated intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge
Clinical improvement of at least one Rutherford classification | baseline, 6, 12, 24 months
  Clinical improvement of at least one Rutherford classification (RCC) compared to pre-procedure RCC
Change in Quality of Life | baseline, 6, 12, and 24 months
  Change in Quality-of-Life Questionnaire (EQ5D) at follow-up, compared to baseline
Limb salvage | 6, 12, 24 months
  Freedom from any above-the-ankle target limb amputation

CONTACTS AND LOCATIONS:
Locations (14):
- Belgium (14):
  - GZA ziekenhuizen, Antwerp, Antwerp
  - UZA, Antwerp, Antwerp
  - Jessa, Hasselt, Limburg
  - CHU Liège, Liège, Liège
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - Vitaz, Sint-Niklaas, Oost-Vlaanderen
  - AZ Sint Jan Brugge, Bruges, West-Vlaanderen
  - O.L.V. Hospital, Aalst
  - Imelda Hospital, Bonheiden
  - A.Z. Sint-Blasius, Dendermonde
  - Z.O.L., Genk
  - az Groeninge, Kortrijk
  - R.Z. Heilig Hart, Tienen
  - A.Z. Jan Portaels, Vilvoorde

IPD SHARING:
Plan to Share IPD: No